CLINICAL TRIAL: NCT02237235
Title: Effect of MMFS-202-302 on Cognitive Enhancement in Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Neurocentria, Inc. (Industry); Brain & Behavior Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00098144
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Results first posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective disorder; Cognition; Magnesium; Imaging; Negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MMFS-202 -302 (Experimental): MMFS-202: evening dose
  MMFS-302: morning dose
  Interventions: Drug: MMFS-202-302
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MMFS-202-302 — Active ingredient: L-Threonic acid Magnesium salt.
  1 g (2 pills) by mouth once daily in the evening for 9 weeks
  Drug: MMFS-302 Active ingredient: L-Threonic Acid Magnesium Salt
  1 g (2 pills) by mouth once daily in the morning for 9 weeks
  Arms: MMFS-202 -302
Drug: Placebo — Two tablets by mouth in the morning, and two tablets by mouth in the evening, daily for 9 weeks.
  Arms: Placebo

SUMMARY:
The goals of this study are to study MMFS-202-302 in a double blind, randomized, placebo-controlled 9-week study of its effect on ameliorating cognitive deficits in 60 patients with schizophrenia or schizoaffective disorder with stable levels of positive symptoms. Secondary end points will include changes in positive and negative symptoms. One dose of MMFS-202-302 will be studied and compared with placebo as adjunctive treatment to atypical antipsychotic drug treatment.

DETAILED DESCRIPTION:
One of the symptoms of schizophrenia is a problem with specific domains of cognition, even when the positive symptoms have been treated. The primary goal of this study is to determine the effectiveness of 9 weeks of supplementation with MMFS-202-302 as augmentation of atypical antipsychotic medication, to improve a critical specific domain of cognitive function, i.e., working memory, in patients with schizophrenia or schizoaffective disorder. To support this primary goal, global function will be assessed with the Clinical Global Impression assessment of change.

The investigators will also examine the effect of MMFS-202-302 on other domains of cognition (e.g. attention, executive function, declarative memory, etc.); negative symptoms of schizophrenia; positive symptoms of schizophrenia; MRI measures of brain structure, resting state functional connectivity, and function during evaluation of emotional/unemotional and rewarding/aversive images and anticipation and receipt of reward and punishment, and working memory; and EEG measurement of network interactivity during learning and memory recollection.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must be capable of giving written informed consent.
2. Male or female subjects of any race; between 18 to 60 years of age, inclusive.
3. No hospitalization other than for evaluation in the past four months
4. Resides in a stable living situation, according to the investigator's judgment.
5. Diagnosis of schizophrenia or schizoaffective disorder of at least one-year duration, as established by the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID-I), and verified with medical records and/or confirmation of diagnosis by the treating clinician. The illness is in a nonacute phase as determined by the subject's primary treating clinician
6. Current psychotropic drug treatment consists of monotherapy with an atypical antipsychotic drug.
7. No more than a mild level of extrapyramidal symptoms (EPS) as determined by the Simpson Angus Scale (SAS) total score: ≤ 6
8. Not taking anticholinergic medication for EPS
9. No evidence of tardive dyskinesia
10. Subjects healthy enough to complete a 9-week clinical trial
11. Women of childbearing potential must have a negative pregnancy test at screening and baseline, and agree to use adequate protection (i.e. double barrier method) for birth control.
12. Able to complete cognition assessments in English
13. General intellectual abilities falling broadly within the average estimated intelligence quotient (IQ) > 80, as measured by the Wide Range Achievement Test - 4th Edition (WRAT-IV).

Exclusion Criteria:

1. Failure to perform screening or baseline examinations
2. Hospitalization within 8 weeks before screening, or change of antipsychotic medication or dose within 2 months prior to screening
3. Subjects who have participated in another clinical trial with an experimental medication within the past 2 months.
4. Patient has had cognitive battery similar to those used in this study within the last 12 months
5. Subjects with other Diagnostic and Statistical Manual (DSM-V) Axis I or Axis II primary diagnoses
6. Diagnosis of alcohol or substance abuse or dependence within the past 3 months,
7. Significant suicide risk as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)
8. Subjects who plan to begin a new course of cognitive remediation therapy, or have been receiving cognitive remediation therapy for less than one year. .
9. History of myocardial infarction, unstable angina, uncontrolled hypotension or hypertension within 3 months before screening.
10. Clinically significant abnormality on screening ECG
11. Alanine transaminase (ALT) or aspartate transaminase (AST) > 2.5 times the upper limit of normal (ULN)
12. History of stroke, brain tumor, head trauma with loss of consciousness, or other clinically significant neurological condition within 12 months before screening
13. Subjects with other uncontrolled medical conditions, in the opinion of the investigator
14. Polypharmacy with two or more antipsychotic drugs or mood stabilizers
15. Use of benzodiazepines
16. Individuals with kidney dysfunction will not be enrolled, as dysfunctional kidneys may have difficulty clearing the magnesium from the body
17. Individuals who are currently taking magnesium supplements

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Y Meltzer, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Psychiatric Clinical Research Program, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MMFS-202 -302: MMFS-202: evening dose
  MMFS-302: morning dose
  MMFS-202-302: Active ingredient: L-Threonic acid Magnesium salt.
  1 g (2 pills) by mouth once daily in the evening for 9 weeks
  Drug: MMFS-302 Active ingredient: L-Threonic Acid Magnesium Salt
  1 g (2 pills) by mouth once daily in the morning for 9 weeks
Period: Overall Study
Arm/Group | MMFS-202 -302 | Placebo
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMFS-202 -302 | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 16 | 29
  White | 12 | 11 | 23
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Matrics Consensus Cognitive Battery (MCCB) [Mean (Standard Deviation); unit: units on a scale] — The Matrics Consensus Cognitive Battery (MCCB) measures cognitive function The MCCB provides an overall composite score, expressed as a T-score, with a mean of 50 and a standard deviation of 10 The MCCB does not have minimum and maximum scores A typical score will fall within a range of 40-60. Scores below 40 indicate impaired cognitive functioning, while scores above 60 suggest above-average cognitive abilities The MCCB is used in clinical research to assess cognitive deficits in individuals with psychiatric disorders, and the T-score scale is used to track cognitive changes over time
  units on a scale | 34.8 (12.6) | 30.8 (12.6) | 32.8 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: MATRICS Consensus Cognitive Battery (MCCB)
Description: Change from Baseline in MATRICS Consensus Cognitive Battery (MCCB) working memory domain.
  The MCCB measures cognitive function. The MCCB provides an overall composite score, expressed as a T-score, with a mean of 50 and a standard deviation of 10 The MCCB does not have minimum and maximum scores due to the use of T scores. A typical score will fall within a range of 40-60. Scores below 40 indicate impaired cognitive functioning, while scores above 60 suggest above-average cognitive abilities.
  The MCCB is often used in clinical research to assess cognitive deficits in individuals with psychiatric disorders, and the T-score scale is used to track cognitive changes over time.
Time Frame: Baseline to Day 63
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MMFS-202 -302 | Placebo
Number analyzed (Participants) | 30 | 30
units on a scale | 41.8 (9.64) | 39.67 (12.86)

2. Secondary Outcome: Overall Clinical Global Impression of Severity Improvement Measured by the Clinical Global Impressions Scale Assessment of Change (CGI-C)
Description: To support the primary endpoint of working memory, the Clinical Global Impression Change (CGI-C) will demonstrate the clinically relevant improvement of global function.
  Minimum is 1 and Maximum is 6. Higher scores means worse outcome.
Time Frame: Day 63
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MMFS-202 -302 | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 3.37 (1.07) | 3.00 (0.95)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | MMFS-202 -302 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 27/30 | 28/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMFS-202 -302 (N=30) | Placebo (N=30)
Headche (Nervous system disorders) | 5 | 4
Insomnia (Psychiatric disorders) | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
pannic attack (Psychiatric disorders) | 0 | 1
blurred vision (Eye disorders) | 0 | 1
Exacerbation of Psychosis (Psychiatric disorders) | 1 | 0
Loose Stool (Gastrointestinal disorders) | 1 | 0
Cutting Self (Psychiatric disorders) | 0 | 1
Stomach ache (Gastrointestinal disorders) | 1 | 1
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (General disorders) | 0 | 2
Hand spasm (Nervous system disorders) | 1 | 0
High triglycerides (Endocrine disorders) | 1 | 0
Shortness of breath (Cardiac disorders) | 0 | 1
Skin Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Flu-like symptoms (Infections and infestations) | 1 | 0
Chest Pressure (Cardiac disorders) | 1 | 0
Diahrrea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 2 | 0
Increase in bowel movements (Gastrointestinal disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
fever (General disorders) | 1 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 1
Strained neck (Musculoskeletal and connective tissue disorders) | 0 | 1
Hospitalization (General disorders) | 0 | 1 — severe in intensity and unrelated to study medication
Drowsiness (General disorders) | 0 | 1
Hospitalization due to diabetic ketoacidosis (Endocrine disorders) | 1 | 0
strep throat (Infections and infestations) | 1 | 0
Hot flashes, sweating, chills (General disorders) | 1 | 0
Dizziness (Light headedness) (Nervous system disorders) | 0 | 1
Pink eye (Eye disorders) | 0 | 1
Nose and chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
dry mouth (General disorders) | 1 | 0
Ingrown toe nail (Musculoskeletal and connective tissue disorders) | 0 | 1
More burping (Gastrointestinal disorders) | 1 | 0
Stomach infection (Gastrointestinal disorders) | 0 | 1
Angioplasty (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT02237235/Prot_SAP_000.pdf